CLINICAL TRIAL: NCT07047638
Title: A Randomized, Evaluator-blinded, No-treatment Controlled, Multicenter Study to Evaluate the Effectiveness and Safety of Restylane Skinboosters Vital Lidocaine for Improvement in Skin Quality of the Face
Brief Title: A Study to Evaluate the Effectiveness and Safety of Restylane Skinboosters Vital Lidocaine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43CH2308
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Skin Quality Improvement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A blind evaluator to assess study primary endpoint.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restylane Skinboosters Vital Lidocaine (Experimental): Subjects in the Treatment Group will be treated with Restylane Skinboosters Vital Lidocaine at Baseline, Week 4 and 8.
  Interventions: Device: Restylane Skinboosters Vital Lidocaine
- No treatment (No Intervention): No treatment control group.

INTERVENTIONS:
Device: Restylane Skinboosters Vital Lidocaine — Restylane Skinboosters Vital Lidocaine is an injectable, sterile, transparent, biodegradable gel of non-animal crosslinked sodium hyaluronate. Restylane Skinboosters Vital Lidocaine has the addition of lidocaine hydrochloride. They are supplied in a glass syringe.
  Arms: Restylane Skinboosters Vital Lidocaine

SUMMARY:
This is a randomized, evaluator-blinded, no-treatment controlled, study to evaluate the effectiveness and safety of Restylane Skinboosters Vital Lidocaine treatment to improve skin quality of the face in China. Subjects of Chinese origin, age 18 years, who are eligible for treatment to improve skin quality of the face. Study center is up to 8.

A total of approximately 171 subjects will be randomized (2:1) to either treatment with Restylane Skinboosters Vital Lidocaine Treatment Group (approximately 114 subjects) or no-treatment Control Group (approximately 57 subjects).

ELIGIBILITY:
Inclusion Criteria:

1. Ability to adequately understand the verbal explanations and the written subject information provided in local language and ability and willingness to give consent to participate in the study. Signed and dated informed consent to participate in the study.
2. Males or non-pregnant, non-breastfeeding females of Chinese origin and 18 years of age or older at the time of signing the Informed Consent Form.
3. Grade 3 (moderate) to 4 (severe) on the 5-grade GSQ-FLS on each side of the face as assessed by the Blinded Evaluator as well as the Treating Investigator (agreement on grade is not required). The GSQ-FLS grade for the right and the left side of the face does not have to be equal.
4. Willing to abstain from any other facial plastic surgical or cosmetic procedures in the face for the duration of the study (e.g., Botulinum toxin, dermal filler, laser or chemical resurfacing, needling, facelift, lifting threads, radiofrequency etc.).
5. Intent to undergo treatment for improvement in skin quality of the face including improvement in fine lines, skin dryness and skin radiance.

   Inclusion criteria 6-7 apply to female subjects only:
6. If the subject is a female of childbearing potential, she agrees to use an acceptable form of effective birth control for the duration of the study and is willing to take a urine pregnancy test (UPT) at screening (or a serum HCG blood test if UPT is not available), Baseline and prior to receiving any study treatment.

   Acceptable forms of effective birth control include:
   * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical caps) with spermicidal foam/gel/film/cream/suppository;
   * Bilateral tubal ligation;
   * Combined oral contraceptives (estrogens and progesterone), implanted or injectable contraceptives on a stable dose for at least 28 days prior to Day 1;
   * Hormonal or copper intra uterine device (IUD) inserted at least 28 days prior to Day 1;
   * Vasectomized partner (in monogamous relationship) for at least 3 months prior to screening;
   * Strict abstinence (at least one month prior to Baseline and agrees to continue for the duration of the study or use acceptable form of birth control).
7. Negative pregnancy test for women of childbearing potential at the screening and Baseline visits.

Exclusion Criteria:

1. Known/previous allergy or hypersensitivity to any injectable hyaluronic acid (HA) gel or to gram positive bacterial proteins.
2. Known/previous allergy or hypersensitivity to anesthetics, e.g., lidocaine or other amide-type anesthetics or nerve blocking agents.
3. Previous or present severe or multiple allergies manifested by severe reactions, such as anaphylaxis or angioedema, or family history of these conditions.
4. Previous facial surgery (e.g., facelift) that in the Treating Investigator´s opinion could interfere with the study safety and/or effectiveness assessments.
5. Any previous aesthetic procedures or implants:

   * Previous permanent filler or implant, lifting threads, or autologous fat in the face regardless of time.
   * Previous use of calcium hydroxylapatite (CaHA), polycaprolactone or poly-L-lactic acid (PLLA) in the treatment area within 24 months.
   * Previous HA filler or collagen filler in the treatment area within 12 months.
   * Previous botulinum toxin treatment in the treatment area within 6 months.
   * Previous energy based aesthetic procedures (e.g., laser, intense pulsed light, radiofrequency, photomodulation and ultrasound) in the treatment area within 6 months.
   * Previous mechanical (e.g., dermabrasion, needling) or chemical aesthetic procedures (e.g., chemical peel) in the treatment area within 6 months.
   * Previous treatment with cryotherapy in the treatment area within 6 months.
6. History of cancer or previous radiation in the treatment area.
7. Advanced photoaged/ photodamaged facial skin (e.g. advanced skin elastosis, multiple lentigo solaris lesions) or skin condition with very crinkled or fragile skin in the face.
8. Presence of any disease or lesions near or on the area to be treated, e.g.:

   * Inflammation, active or chronic infection (e.g., in mouth, dentals, head, eye);
   * Current cutaneous inflammatory or infectious processes near or on the area to be treated (e.g., acne, dermatitis, herpes) which, in the Treating Investigator's opinion, would interfere with the study injections and/or study assessments;
   * Scars (other than from acne) or deformities;
   * Cancer, or precancerous conditions (e.g., actinic keratosis or actinic cheilitis).
9. Evidence of scar-related disease or delayed healing activity within 1 year prior to the Baseline visit, or subjects susceptible to keloid formation, hyperpigmentation or hypertrophic scarring in the opinion of the Investigator.
10. Presence of tattoo, piercing, beard or facial hair, which, in the Treating Investigator's opinion, would interfere with the study injections and/or study assessment.
11. Presence of a dental, oral, or facial condition which, in the Treating Investigator's opinion, would interfere with the study injections and/or study assessments, e.g., has dentures or any device covering all or part of the upper palate, and/or severe malocclusion or dentofacial or maxillofacial deformities. Any planned procedure (e.g., dental implants, tooth extractions, orthodontia) during the study period, that would make the subject unsuitable for inclusion in the opinion of the Investigator.
12. An underlying known disease, a surgical or medical condition that would expose the subject to undue risk, e.g., history of bleeding disorders, active hepatitis, active autoimmune disease such as connective tissue diseases, systemic lupus erythematosus, polymyositis, dermatomyositis, or scleroderma.
13. Use of concomitant medication that have the potential to prolong bleeding times such as anticoagulants or inhibitors of platelet aggregation (e.g., warfarin, clopidogrel, aspirin or other non-steroidal anti-inflammatory drugs [NSAIDs], Omega-3 or Vitamin E), within 14 days prior to injection. Omega-3 and Vitamin E are acceptable only as part of a standard multivitamin formulation. Cyclooxygenase-2 (COX 2) inhibitors are allowed.
14. Treatment with chemotherapy, immunosuppressive agents, systemic corticosteroids within 3 months before treatment (eyedrops, intraarticular, and inhaled corticosteroids are allowed).
15. Use of topical corticosteroids or prescription retinoids on the treatment area within 1 months prior to Baseline or use of systemic retinoids within 6 months prior to Baseline.
16. Presence of any condition or situation, which in the opinion of the Treating Investigator makes the subject unable to complete the study per protocol, e.g.

    * Subject is not likely to avoid other prohibited facial cosmetic treatments;
    * Subject is not likely to complete the study because of other commitments;
    * Subject is anticipated to be unavailable for visits, incapable of understanding the investigational assessments or having unrealistic expectations of treatment result;
    * Subject who has a concomitant condition (e.g., acute viral or bacterial infection with fever) that might confuse or confound study treatments or assessments.
17. Study center personnel, close relatives of the study center personnel (e.g., parents, children, siblings, or spouse), employees or close relatives of employees at the Sponsor company.
18. Participation in any other interventional clinical study within 30 days before treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Responder rate based on the Blinded Evaluators' live assessment using the Galderma Skin Quality - Fine Lines Scale (GSQ-FLS). | At Week 12 after Baseline
  A responder is defined as a subject with at least 1-grade improvement from Baseline in both sides of the face concurrently on the scale. GSQ-FLS is a 5-grade scale with a higher score meaning a worse situation in fine line.

SECONDARY OUTCOMES:
Responder rate based on the Blinded Evaluators' live assessment using the GSQ-FLS | At Week 16, 20, 24, 36, 48 and 60 after Baseline for the Treatment Group or at Week 16, 20 and 24 after Baseline for the no-treatment Control Group. GSQ-FLS is a 5-grade scale with a higher score meaning a worse situation in fine line.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China